CLINICAL TRIAL: NCT04603443
Title: Supplementation With Amino Acid Rehabilitative Therapy in TBI (SmART-TBI): A Randomized Placebo-Controlled Trial to Improve Sleep
Brief Title: SmART-TBI: Supplementation With Amino Acid Rehabilitative Therapy in TBI
Acronym: SmART-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Children's Hospital of Philadelphia (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURR-003-19F; I01CX002022 (NIH)
Record Dates: First submitted 2020-10-02; First posted 2020-10-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; sleep; cognition; bcaa
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled feasibility study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and study team members will be double blinded to intervention. The biostatistician and Research Pharmacist dispensing drug will be the only ones with the key to unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BCAA 20g/daily (Experimental): Branched Chain Amino Acids, 10g BID x 12 weeks
  Interventions: Dietary Supplement: Branched Chain Amino Acids
- BCAA 40g/daily (Experimental): Branched Chain Amino Acids, 20g BID x 12 weeks
  Interventions: Dietary Supplement: Branched Chain Amino Acids
- BCAA 60g/daily (Experimental): Branched Chain Amino Acids, 30g BID x 12 weeks
  Interventions: Dietary Supplement: Branched Chain Amino Acids
- Placebo 20g/daily (Placebo Comparator): Protein without BCAA, 10g BID x 12 weeks
  Interventions: Dietary Supplement: Protein Control

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acids — Isoleucine, Leucine, and Valine, 10g BID x 12 weeks
  Other Names: BCAA-20
  Arms: BCAA 20g/daily
Dietary Supplement: Branched Chain Amino Acids — Isoleucine, Leucine, and Valine, 20g BID x 12 weeks
  Other Names: BCAA-40
  Arms: BCAA 40g/daily
Dietary Supplement: Branched Chain Amino Acids — Isoleucine, Leucine, and Valine, 30g BID x 12 weeks
  Other Names: BCAA-60
  Arms: BCAA 60g/daily
Dietary Supplement: Protein Control — Protein placebo control - all amino acids except for BCAA, 10g BID x 12 weeks
  Arms: Placebo 20g/daily

SUMMARY:
The most persistent and disabling postconcussive symptoms following mild traumatic brain injury (mTBI) are sleep disturbances and cognitive dysfunction, with few tractable interventions currently available. Here, a novel therapy will be tested consisting of dietary supplementation with branched chain amino acids (BCAA), based on the study team's previous preclinical work showing restoration of glutamate neurotransmitter balance in sleep and memory circuits. Supplementation with Amino acid Rehabilitative Therapy in TBI (SmART-TBI) is a randomized, placebo-controlled, double-blinded, exploratory clinical trial of BCAA intended to establish the feasibility, acceptability, and limited efficacy of long-term BCAA to improve sleep and cognition in Veterans with mTBI. These results will inform the optimal study design of a future, full-scale randomized controlled trial, including the identification of the proper dose and duration of BCAA to improve sleep and the potential subpopulations of Veterans with mTBI that may benefit the most.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI) has impacted over 60% of all OEF/OIF Veterans over the past decade, and over 20% of these Veterans carry a diagnosis of postconcussion syndrome. Arguably the most disabling postconcussion symptoms are sleep-wake and cognitive disturbances. Sleep, cognitive function, and related symptoms often remain impaired >10-15 years following mTBI. Not only are these symptoms themselves exceedingly difficult to live with, but poor sleep and cognition also interfere with ongoing rehabilitation interventions, and prevent reintegration into civilian life and return to gainful employment. Most existing therapies for sleep-wake and cognitive dysfunction following mTBI are merely symptomatic, and they also suffer from low efficacy and/or patient acceptability. Thus, there is an urgent need to identify mechanism-based interventions for sleep and cognitive problems following mTBI, in order to facilitate optimal rehabilitation and functional outcomes.

The study team's long-term goal is to implement a brain-bioactive pharmacological intervention to address sleep and cognitive disturbance in individuals with mTBI. The overall objective of this application, which represents the first step towards this goal, is to test the feasibility and limited efficacy of a highly promising therapy consisting of a dietary supplement, branched chain amino acids (BCAA; i.e., leucine, isoleucine, and valine), to treat sleep disturbances in individuals with mTBI. There is compelling scientific precedent and safety data to support the testing of BCAA therapy in Veterans with mTBI. Preliminary preclinical data has shown that the mechanism of action for BCAA, acting as a precursor to the excitatory neurotransmitter glutamate, restores the balance of excitation to inhibition within the dysfunctional brain circuits for both sleep and cognition in mTBI. With these data, the study team has also meticulously mapped the optimal dosing, duration, and route of administration in mice. Further, the study team now has pilot data from a double-blinded, placebo-controlled study showing that 3 weeks of dietary BCAA supplementation, but not placebo, significantly improved self-reported sleep in Veterans. Other research groups have used dietary BCAA supplementation in humans across multiple conditions at doses up to 60 grams/day and durations up to 12 months with few to no side effects.

The central hypothesis is that BCAA dietary supplementation will improve sleep quality in Veterans with mTBI. As a first step towards testing this hypothesis, herein is proposed a long-term feasibility, acceptability, and limited efficacy study of BCAA's effects on sleep that will be randomized, placebo-controlled, and double-blinded. Veterans with mTBI will be randomly assigned to receive BCAA at 20, 40 or 60 grams/day per oral (PO) or a placebo (n=50 per group) for 12 weeks. Feasibility, acceptability, and limited efficacy outcomes based on sleep (e.g., self-report, continuous actigraphy, and overnight polysomnography) will be assessed.

Results will inform the optimal study methodology and design for a future, full-scale randomized controlled trial, including the identification of the proper dose and duration of BCAA to improve sleep and the potential subpopulations of Veterans with mTBI that may be differentially affected by BCAA. This work will aos be used to generate hypotheses on the effect of BCAA on cognition and overall quality of life measures to inform future research.

ELIGIBILITY:
Inclusion Criteria:

* Be Veterans (male and female; any race; 18-65 years of age)
* Be English speaking
* Be accessible via phone
* Be non-decisionally impaired
* Attest to there being no chance of being or becoming pregnant during the study (if female)
* Attest to no history of maple syrup urine disease or known family history of maple urine syrup disease
* Have either a history of self-reported sleep disturbances, either as determined via the Insomnia Severity Index, Functional Outcomes of Sleep Questionnaire or Epworth Sleepiness Scale, clinical assessment, and/or a history of self-reported cognitive disturbance (e.g., poor memory, concentration, attention)
* Not have an allergy to sucralose
* Not be a shift worker (e.g. have worked night or rotating shifts more than twice in the past month)
* Not have a diagnosis of amyotrophic lateral sclerosis
* Not be currently supplementing their diet with branched chain amino acids
* Not be starting another sleep intervention (e.g., positive airway pressure therapy for sleep apnea, sedative-hypnotic medication, or cognitive behavioral therapy for insomnia) during the study

  * if already engaged in another sleep intervention, this must be stable and not undergo further changes during the study
* Meet diagnostic criteria for TBI using a validated clinical interview

Exclusion Criteria:

* Pregnancy or female trying to conceive
* Under 18 years old
* Known history of maple syrup urine disease
* Dementia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Actiwatch Adherence | Year 1
  Proportion of days with actiwatch worn (goal >70% days)
Study Drug Adherence by drug accounting | Year 1
  Proportion of study drug consumed within each timepoint assessed by drug accounting.
Study drug adherence by sleep diary | Year 1
  Proportion of study drug consumed assessed by sleep diary.
Change in Monitoring of Side Effects Scale (MOSES) | 12 weeks
  Change in Monitoring of side effects scale with emphasis on GI, neurological, psychiatric side effects. Range= 0-124, higher= more side effects.
Study Drug Adherence by serum or sweat assay | Year 1
  Proportion of study drug consumed assessed by serum or sweat assays of BCAA (goal >70% and >20% increase in levels.
Patient satisfaction with overall study process | 12 weeks
  Likert scale (1-5, higher= more satisfied) assessing satisfaction with consent process, staff, medication dispensing and regimen, devices/equipment, sleep study, questionnaires, cognitive testing, and overall experience of the study.
Monitoring of Side Effects Scale (MOSES) | 4 weeks
  Monitoring of side effects scale with emphasis on GI, neurological, psychiatric side effects. Range= 0-124, higher= more side effects.
Change in Monitoring of Side Effects Scale (MOSES) | 8 weeks
  Change in Monitoring of side effects scale with emphasis on GI, neurological, psychiatric side effects. Range= 0-124, higher= more side effects.
Reasons for non-adherence | 4 weeks
  Likert scale questions assessing response to statements including: "It upset my stomach", "I didn't have time", "it was too much to drink", "I didn't like the taste", "I didn't feel a benefit". Scale= 0-25, higher=agree more with statement.
Change in Reasons for non-adherence | 8 weeks
  Change in Likert scale questions assessing response to statements including: "It upset my stomach", "I didn't have time", "it was too much to drink", "I didn't like the taste", "I didn't feel a benefit". Scale= 0-25, higher=agree more with statement.
Change in Reasons for non-adherence | 12 weeks
  Change in Likert scale questions assessing response to statements including: "It upset my stomach", "I didn't have time", "it was too much to drink", "I didn't like the taste", "I didn't feel a benefit". Scale= 0-25, higher=agree more with statement.
Recruitment | Year 1
  Number of subjects consented of those eligible as descriptive percent
Recruitment source | Year 1
  Proportion of subjects recruited from various sources (clinical referral, flyers, ads, etc)
Retention | Year 1
  Number of completers out of the total number consented as descriptive statistic
Retention by arm | Year 1
  Proportion of drop out within each arm
Incidence of non-participation | Year 1
  Reasons for not participating after initial contact and before consent as descriptive percent.
Screen Failures | Year 1
  Number of subjects enrolled who were later found ineligible as a descriptive percent
Screen Failures | Year 2
  Number of subjects enrolled who were later found ineligible as a descriptive percent
Screen Failures | Year 3
  Number of subjects enrolled who were later found ineligible as a descriptive percent
Screen Failures | Year 4
  Number of subjects enrolled who were later found ineligible as a descriptive percent
Incidence of non-participation | Year 2
  Reasons for not participating after initial contact and before consent as descriptive percent.
Incidence of non-participation | Year 3
  Reasons for not participating after initial contact and before consent as descriptive percent.
Incidence of non-participation | Year 4
  Reasons for not participating after initial contact and before consent as descriptive percent.
Retention by arm | Year 2
  Proportion of drop out within each arm
Retention by arm | Year 3
  Proportion of drop out within each arm
Retention by arm | Year 4
  Proportion of drop out within each arm
Retention | Year 2
  Number of completers out of the total number consented as descriptive statistic
Retention | Year 3
  Number of completers out of the total number consented as descriptive statistic
Retention | Year 4
  Number of completers out of the total number consented as descriptive statistic
Recruitment source | Year 2
  Proportion of subjects recruited from various sources (clinical referral, flyers, ads, etc)
Recruitment source | Year 3
  Proportion of subjects recruited from various sources (clinical referral, flyers, ads, etc)
Recruitment source | Year 4
  Proportion of subjects recruited from various sources (clinical referral, flyers, ads, etc)
Recruitment | Year 2
  Number of subjects consented of those eligible as descriptive percent
Recruitment | Year 3
  Number of subjects consented of those eligible as descriptive percent
Recruitment | Year 4
  Number of subjects consented of those eligible as descriptive percent
Study Drug Adherence by serum or sweat assay | Year 2
  Proportion of study drug consumed assessed by serum or sweat assays of BCAA (goal >70% and >20% increase in levels.
Study drug adherence by serum or sweat assay | Year 3
  Proportion of study drug consumed assessed by serum or sweat assays of BCAA (goal >70% and >20% increase in levels.
Study drug adherence by serum or sweat assay | Year 4
  Proportion of study drug consumed assessed by serum or sweat assays of BCAA (goal >70% and >20% increase in levels.
Study Drug Adherence by sleep diary | Year 2
  Proportion of study drug consumed assessed by sleep diary.
Study Drug Adherence by sleep diary | Year 3
  Proportion of study drug consumed assessed by sleep diary.
Study Drug Adherence by sleep diary | Year 4
  Proportion of study drug consumed assessed by sleep diary.
Study drug adherence by drug accounting | Year 2
  Proportion of study drug consumed within each timepoint assessed by drug accounting.
Study drug adherence by drug accounting | Year 3
  Proportion of study drug consumed within each timepoint assessed by drug accounting.
Study drug adherence by drug accounting | Year 4
  Proportion of study drug consumed within each timepoint assessed by drug accounting.
Actiwatch Adherence | Year 2
  Proportion of days with actiwatch worn (goal >70% days)
Actiwatch Adherence | Year 3
  Proportion of days with actiwatch worn (goal >70% days)
Actiwatch Adherence | Year 4
  Proportion of days with actiwatch worn (goal >70% days)

CONTACTS AND LOCATIONS:
Overall Officials: Miranda M Lim, MD PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying any individual whose data are included in the dataset.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after the resulting publication
Access Criteria: Final datasets will be maintained locally until institutional resources become available for public access to data sets. Limited de-identified data sets will be made available on a case-by-case basis in response to specific user requests that meet criteria specified above.

DOCUMENTS (1):
  • Informed Consent Form (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT04603443/ICF_000.pdf